CLINICAL TRIAL: NCT04571047
Title: Time to Surgery - the Impact of Waiting Time on Outcome After Colorectal Cancer Treatment
Acronym: Tidop
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor of surgery, Sahlgrenska University Hospital
Other Study IDs: Tidop
Record Dates: First submitted 2020-09-02; First posted 2020-09-30 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Time-to-Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Patients diagnosed with colonrectal cancer between 2008-2016
  Interventions: Other: Time to treatment

INTERVENTIONS:
Other: Time to treatment — Treatment before or after 4 weeks after diagnosis

SUMMARY:
We aim to perform a register-based, observational cohort study to investigate whether it is safe to delay start of treatment with a curative intention after a colorectal cancer diagnosis. Our hypothesis is that delaying start of treatment until 4-8 weeks is as safe as starting treatment within four weeks after a colorectal cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colorectal cancer 2008-2016 in Sweden

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients registered with a diagnosis of colorectal cancer in Sweden between 2008-2016
Sampling Method: Probability Sample
Enrollment: 40000 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Overall survival

SECONDARY OUTCOMES:
Length of stay | 90 days
  Hospital stay
Re-operations within 3 months | 90 days
  Surgical procedures registered within 3 months after the procedure date
Re-admissions within 3 months | 90 days
  Readmissions registered within 3 months after the procedure date
Radical surgery | 90 days
  Defined as R0 resection

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, Principal Investigator — Sahlgrenska Universitetssjukhuset
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The data is extracted from CRCBaSe, (ColoRectal Cancer Data Base) a combination of several registries in Sweden and thus the sharing option will be decided by that work group